CLINICAL TRIAL: NCT01529164
Title: Phase II Study of Recombinant Endostatin Combined With Modified FOLFOX6 in Advanced Colorectal Cancer
Brief Title: Efficacy and Safety Study of Recombinant Endostatin Combined With Chemotherapy to Treat Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Simcere Pharmaceutical Co., Ltd (Other)
Responsible Party: Principal Investigator, Lin Yang, associated professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-023
Record Dates: First submitted 2012-02-04; First posted 2012-02-08 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Colorectal Cancer
Keywords: endostatin; chemotherapy; antiangiogenesis agent; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Endostatins; endostar protein; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Experimental)
  Interventions: Drug: Endostatins (Endostar); Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-fluorouracil

INTERVENTIONS:
Drug: Endostatins (Endostar) — 7.5mg/m2 iv d1-10,repeat every 14 days,until progression or occurrence of untolerated toxicity
  Other Names: Endostar
Drug: Oxaliplatin — 85mg/m2 iv d1 ,repeat every 14 days,until progression or occurrence of untolerated toxicity
  Other Names: Eloxatin
Drug: Leucovorin — 200mg/m2 iv d1 ,repeat every 14 days
Drug: 5-fluorouracil — 400mg/m2 iv bolus,then 2400mg/m2 continuous infusion for 46 hours,repeated every 14 days,until progression or occurrence of untolerated toxicity

SUMMARY:
Studies suggest that the addition of antiangiogenic agents to conventional therapeutic strategies, e.g., chemotherapy, radiation, or other tumor-targeting agents, will increase clinical efficacy. For advanced colorectal cancer,the antiangiogenic agent bevacizumab has become an important treatment option and its combination with chemotherapy is now being one of the standard first line therapy. This phase II study was conducted to determine the efficacy and safety of another antiangiogenesis inhibitor rh-endostatin plus mFOLFOX6 in advanced colorectal cancer.

DETAILED DESCRIPTION:
Rh-Endostatin (Endostar; Simcere Pharmaceutical Co., Ltd, JiangSu,China) is a humanized recombinant endostatin which is a direct angiogenesis inhibitor targeting the microvascular endothelial cells (ECs). A pivotal phase III study completed in China demonstrated that the addition of rh-endostatin to navelbine plus cisplatin conferred clinically significant improvements in overall survival (OS), progression-free survival (PFS), as well as response rate (RR), in patients with previously untreated metastatic non small cell lung cancer (NSCLC). In vitro, the combination of Endostatin and fluorouracil showed synergistic activity in inhibiting colon cancer. MFolfox6 was standard first-line regimen in advanced colorectal cancer. The investigators carried out a phase II trial to investigate the activity and safety of rh-endostatin plus mFOLFOX in patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent (IC)
* Age greater than or equal to 18 years
* Histologically or cytologically confirmed metastatic or recurrent colorectal tumors with no previous treatment for advanced disease.
* At least one measurable lesion according to the RECIST criteria which has not been irradiated (i.e. newly arising lesions in previously irradiated areas are accepted). Minimum indicator lesion size: > 10 mm measured by spiral CT or >20mm measured by conventional techniques
* ECOG performance status 0-1
* Life expectancy > 3 months
* ECG is normal

Exclusion Criteria:

* Pregnant or lactating woman
* Any prior oxaliplatin treatment, with the exception of adjuvant therapy given > 12 months prior to the beginning of study therapy,and any prior 5-fluorouracil treatment, with the exception of adjuvant therapy given > 6 months prior to the beginning of study therapy
* Any prior endostatin treatment
* known hypersensitivity to 5-fluorouracil,oxaliplatin,leucovorin
* History of persistent neurosensory disorder including but not limited to peripheral neuropathy
* known DPD deficiency
* Treatment for other carcinomas within the last five years, except cured non-melanoma skin and treated in-situ cervical cancer
* Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) within the last 6 months
* Any of the following laboratory values:

  * Abnormal hematologic values (neutrophils < 1.5 x 109/L, platelet count < 100 x 109/L)
  * Urine protein: creatinine ratio >/= 1.0, Impaired renal function with estimated creatinine clearance < 30 ml/min
  * Serum bilirubin > 1.5 x upper normal limit. ALT, AST > 2.5 x upper normal limit (or > 5 x upper normal limit in the case of liver metastases)
  * Alkaline phosphatase > 2.5 x upper normal limit (or > 5 x upper normal limit in the case of liver metastases or > 10 x upper normal limit in the case of bone disease)
* use of full-dose anticoagulants or thrombolytics
* known CNS metastases
* serious nonhealing wound, ulcer, or bone fracture
* clinically significant bleeding diathesis or coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
response rate | 3 years
  From date of treatment was administered until the date of first documented response according to RECIST criteria

SECONDARY OUTCOMES:
progression free survival | 3 years
  From date of chemotherapy was administered until the date of first documented progression or date of death from any cause, whichever came first, assessed every 8 weeks.
overall survival | 3 years
  From date of treatment was administered until the date of death from any cause, assessed every 3 months.
Number of participants with adverse events | 3 years
  assessed from the date of treatment to 1 month after stop treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lin Yang, MD, Principal Investigator — Cancer hospital&institute,Chinese Academy of Medical Sciences
Locations (1):
- Cancer hospital & Institute,Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China